CLINICAL TRIAL: NCT01018576
Title: Delayed Cord Clamping: Prevention of Anemia and Hypothermia in Premature Infants
Brief Title: Delayed Cord Clamping in Premature Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate numbers of babies enrolled and departure of co-investigator
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 200916964
Record Dates: First submitted 2009-11-05; First posted 2009-11-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Hypothermia; Anemia
Keywords: delayed cord clamping; premature infants; hypothermia; anemia; intraventricular hemorrhage; Anemia in premature infants
MeSH Terms: conditions — Hypothermia; Anemia; Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Delayed cord clamping (Experimental)
  Interventions: Other: Delayed cord clamping

INTERVENTIONS:
Other: Delayed cord clamping — Infants will be covered with plastic and placed on a chemical warmer at delivery and then clamping of the umbilical cord will be delayed for 30-60 seconds.

SUMMARY:
Delayed cord clamping has been shown to decrease the risk of bleeding in the brain of premature infants. However this procedure is not standard due to concerns that the premature infant will get too cold. In this study the investigators look at using a plastic covering and a chemical warmer to keep the small premature baby warm while waiting 30-60 seconds to clamp the umbilical cord.

DETAILED DESCRIPTION:
Enrolled premature infants will be compared to age matched historical controls that did not receive delayed cord clamping but were placed under a warmer immediately after birth. Outcomes to be analyzed include initial body temperature, hematocrit at birth and 24 hours of age, number of red blood cell transfusions during hospital stay, umbilical cord gas, first blood gas following delivery, blood pressure data in the first 24 hours, fluid bolus and inotrope requirement in the first 24 hours, incidence of intraventricular hemorrhage and late-onset sepsis, peak bilirubin level, length of phototherapy, and Apgar scores.

ELIGIBILITY:
Inclusion Criteria:

* premature infants at 24-28 completed weeks gestation at the time of delivery
* informed consent obtained from parents prior to delivery

Exclusion Criteria:

* multiple gestation (twins, triplets, etc)
* prolonged fetal bradycardia
* placental abruption or previa
* maternal illness
* major congenital anomalies
* maternal fever in labor
* fetal illness (e.g. isoimmune hemolysis)

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Initial body temperature | At birth

SECONDARY OUTCOMES:
Hematocrit at birth and 24 hours of age | first day of life

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Underwood, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States